CLINICAL TRIAL: NCT04344834
Title: Psychological Impact of Covid-19 on The Egyptians
Brief Title: Short and Long-term Psychological Impact of Covid-19 on The Egyptians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, Lecturer of Psychiatry, Assiut University
Other Study IDs: Covid-19 mental health
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Mental Health Issue
Keywords: Covid-19; Egyptian; Health workers; population; mental health
MeSH Terms: conditions — COVID-19; Psychological Well-Being | interventions — Tooth Exfoliation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health care workers: Egyptian health care workers
  Interventions: Diagnostic Test: A questionnaire or scales
- General population: Any Egyptian personnel
  Interventions: Diagnostic Test: A questionnaire or scales
- Recovered fromCOVID-19: Patients recovered from COVID-19
  Interventions: Diagnostic Test: A questionnaire or scales

INTERVENTIONS:
Diagnostic Test: A questionnaire or scales — A questionnaire or scale to assess the participants mental health.

SUMMARY:
The World Health Organization (WHO) has recently declared coronavirus disease 2019 (Covid-19) a public health emergency of international concern. Impact of the pandemic of covid-19 on the mental health of patients, health care workers and general population would be affected.

DETAILED DESCRIPTION:
Health care workers and general population will be included in the study. A questionnaire will be used to assess their knowledge and practices regarding covid-19 and its impact on mental health.

Patients Mental health will be assessed regarding anxiety, depression and obsessive compulsive disorder, sleep disorder will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian population

Exclusion Criteria:

* Patients not accepting to participate in the questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health care workers, patients recovered from COVID-19 and general population
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression | 6 months
  Hamilton depression scale:The total score is obtained by summing the score of each item, 0-4 (symptom is absent, mild, moderate, or severe). For the 17-item version, scores can range from 0 to 54.Where total scores between 0 and 7 do not indicate the presence of depression, scores between 8 and 13 indicate mild depression, scores between 14 and 18 indicate moderate depression, scores between 19 and 22 indicate severe depression and 23 score or more indicate very severe depression.
Anxiety | 6 months
  Hamilton anxiety scale:The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where total score 0 -13=normal, 14-17 = mild anxiety, 18-24 = moderate anxiety, 25-30 = severe anxiety.
Obsessive compulsive disorder | 6 months
  Yale-Brown Obsessive Compulsive Scale (OCD): Each item is rated from 0 (no symptoms) to 4 (extreme symptoms). A score of 0-7 is considered nonclinical. Scores ranging between 8 and 15 are considered mild. Scores between 16 and 23 are considered moderate and scores between 24-31 and 32-40 are considered severe and extreme, respectively.
Sleep disorder | 6 months
  Pitsburgh sleep quality index
Psychological problems | 6 months
  Symptom checklist 90

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Only the data described in the results of the study.